CLINICAL TRIAL: NCT05990374
Title: Therapeutic Effects and Effects on Body Fat of GLP-1 Receptor Agonists in Patients With Type 2 Diabetes for 1-4 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20220825-04
Record Dates: First submitted 2023-07-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dulaglutide (Active Comparator): Once a week, subcutaneous injection
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc
- semaglutide (Active Comparator): Once a week, subcutaneous injection
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc
- Loseenatide (Active Comparator): Once a week, subcutaneous injection
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc
- tirzepatide (Active Comparator): Once a week, subcutaneous injection
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc
- elbenatide (Active Comparator): Once a week, subcutaneous injection
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc
- original treatment (Active Comparator): Once a week, subcutaneous injection
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc
- placebo (Placebo Comparator): The patients will be treated according to the original protocol
  Interventions: Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc

INTERVENTIONS:
Drug: Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc — The study compared patients taking different types of GLP-1(Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc) with taking placebo.

SUMMARY:
The efficacy of long-term treatment with different GLP-1RA (Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc.) was evaluated through 1-4 years of follow-up, and the effects of long-term treatment on blood glucose and body fat of patients.

DETAILED DESCRIPTION:
At present, there has been no evaluation on the efficacy of long-term treatment of different GLP-1RA (Duragtide, Semaglutide, losenatide, tirzepatide, ebenatide, etc.), and the effects of long-term treatment on patients' blood glucose and body fat. This study intends to follow up for 1-4 years. To observe the effects of different GLP-1RA on body fat, insulin resistance, body weight, blood glucose, blood lipids, stomach volume, etc., in patients with type 2 diabetes, and explore the factors affecting the efficacy, so as to provide more evidence-based medical evidence for drug treatment and benefit patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type 2 diabetes according to the 1999 WHO standards;
2. received at least 8 weeks of simple diet control and physical exercise before screening; Patients with type 2 diabetes who were treated with stable hypoglycemic drugs and had inadequate glycemic control within 8 weeks prior to screening;
3. HbA1c≥7.5%；
4. BMI>24kg/m2;
5. Subjects agree to maintain a scientific diet and exercise habits throughout the study, and regularly self-monitor and record blood sugar (SMBG);
6. Be willing to sign written informed consent and comply with the study protocol

Exclusion Criteria:

1. Use of any of the following drugs or treatments in the 3 months prior to screening: treatment with GLP-1RA, GLP-1 analogue, DPP-4 inhibitor, or any other incretin analogue;
2. Long-term (more than 7 consecutive days) intravenous administration, oral administration, or intra-articular administration of corticosteroids within 2 months prior to screening;
3. Use of weight control drugs or surgery that can lead to weight instability within 2 months before screening, or are currently in a weight loss program and not in the maintenance stage:
4. History of acute and chronic pancreatitis; A history of medullary C-cell carcinoma, MEN (multiple endocrine tumors) 2A or 2B syndrome, or related family history;
5. Clinically significant gastric emptying abnormalities;
6. tumors of any organ system that have been treated or not treated in the 5 years prior to screening;
7. had received coronary angioplasty, coronary stenting, or coronary artery bypass within 6 months before screening. Negligent compensatory heart failure (NYHA rating III and IV), stroke or transient ischemic attack, unstable angina, myocardial infarction, persistent and clinically significant arrhythmia;
8. Acute metabolic complications occurred within 6 months before screening;
9. Before screening, any of the laboratory test indicators meet the following criteria: glutamic-pyrugenic transaminase >2.5 times or ASpartate transaminase >2.5 times; eGFR <45ml/min/1.73m2; Fasting glycerin tricol >5.64mmol/L.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Effects of different GLP-1 on blood glucose | 1,2,3,4 year
  The changes of blood glucose fluctuation after treatment

SECONDARY OUTCOMES:
Effects of different GLP-1 on body fat mass | 1,2,3,4 year
  The changes of body fat mass after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical Univesity, Nanjing, China

REFERENCES:
- [Derived] Xu CL, Kong XC, Liu XM, Xu XH, Liu BL, Ma JH. Effect of Ebenatide on glycemic metabolism and body fat in patients with type 2 diabetes mellitus. Front Endocrinol (Lausanne). 2025 Jun 18;16:1622526. doi: 10.3389/fendo.2025.1622526. eCollection 2025. PMID 40607222